CLINICAL TRIAL: NCT05735431
Title: Phase 3, Multicenter, Randomized, Parallel-Group, Open-Label, Comparative Non-Inferiority Fixed-Dose Combination Formoterol 6 mcg/Fluticasone 125 mcg Versus Alenia® (Formoterol 6 mcg/Budesonide 200 mcg) in the Treatment of Moderate Asthma
Brief Title: Non-Inferiority,Combination Formoterol/FluticasonexAlenia®Formoterol/Budesonide for Asthma in Brazil
Acronym: FORASMA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic change in development priorities
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF182
Record Dates: First submitted 2022-12-13; First posted 2023-02-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Moderate Asthma
MeSH Terms: interventions — Formoterol Fumarate; Fluticasone

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized to one of the following treatment groups:
  Investigational Group: Formoterol 6 mcg/fluticasone 125 mcg Eurofarma. Participants randomized to this group will receive 1 inhalation of the product, twice daily, for 12 weeks.
  Comparator Group: Alenia® 6 mcg/200 mcg. Participants randomized to this group will receive 1 inhalation of the product, twice daily, for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formoterol 6 mcg/fluticasone 125 mcg (Experimental): Formoterol 6 mcg/fluticasone 125 mcg Eurofarma.
  Interventions: Drug: Administration of investigation drug
- Alenia® 6 mcg/200 mcg (Active Comparator): Alenia® 6 mcg/200 mcg.
  Interventions: Drug: Administration of comparator

INTERVENTIONS:
Drug: Administration of investigation drug — Participants randomized to this group will receive 1 inhalation of the product, twice daily, for 12 weeks.
  Other Names: Formoterol 6 mcg/fluticasone 125 mcg
  Arms: Formoterol 6 mcg/fluticasone 125 mcg
Drug: Administration of comparator — Participants randomized to this group will receive 1 inhalation of the product, twice daily, for 12 weeks.
  Other Names: Alenia® 6 mcg/200 mcg
  Arms: Alenia® 6 mcg/200 mcg

SUMMARY:
Eurofarma Laboratórios S.A. markets a FDC containing formoterol 12 mcg/fluticasone 250 mcg, in a single capsule for inhalation (Lugano®; reference product). The product is indicated for the treatment of asthma in patients aged ≥ 12 years. The company seeks to register a product with lower concentrations of mono-drugs (6 mcg and 125 mcg, respectively) to enable the dosage step up and step down treatment strategies advocated by the Global Initiative for Asthma for the inhaled maintenance treatment of asthma (GINA, 2022 ) with these combinations.

This Phase 3 study will be carried out for demonstrating the non-inferiority of the investigational drug (FDC of formoterol 6 mcg/fluticasone 125 mcg) compared to the FDC of formoterol 6 mcg/budesonide 200 mcg (Alenia® - Aché Laboratórios Farmacêuticos S.A.) in the maintenance treatment of asthma, allowing its registration as a new concentration of the drug already registered by the company.

DETAILED DESCRIPTION:
The investigational drug consists of a fixed-dose combination (FDC) that contains formoterol fumarate dihydrate , a long-acting β2-agonist (LABA), and fluticasone propionate , a glucocorticoid, powder for inhalation contained in a single capsule, in concentrations of 6 mcg and 125 mcg per capsule, respectively. The investigational drug consists of a fixed-dose combination (FDC) that contains formoterol fumarate dihydrate , a long-acting β2-agonist (LABA), and fluticasone propionate , a glucocorticoid, powder for inhalation contained in a single capsule, in concentrations of 6 mcg and 125 mcg per capsule, respectively.The investigational drug consists of a fixed-dose combination (FDC) that contains formoterol fumarate dihydrate , a long-acting β2-agonist (LABA), and fluticasone propionate , a glucocorticoid, powder for inhalation contained in a single capsule, in concentrations of 6 mcg and 125 mcg per capsule, respectively. Multicenter, randomized, parallel-group, open-label, comparative non-inferiority clinical trial. After a run-in period of four (04) weeks, during which all participants will receive Alenia® 6 mcg/200 mcg, patients with moderate asthma (step 3) controlled according to the criteria of the Global Initiative for Asthma (GINA, 20221) will be randomized in a 1:1 ratio to receive the FDC of formoterol 6 mcg/fluticasone 125 mcg Eurofarma (investigational drug) or Alenia® 6 mcg/200 mcg (comparator drug) (one [01] inhalation, twice a day) for 12 weeks. The primary non-inferiority assessment will be performed at the end of the 12 weeks of treatment. 2The study will be conducted in an open-label scenario, since the inhalation devices for the products have different aspects, making it impossible to blind the study treatments. The objective nature of the primary efficacy variable (forced expiratory volume in one second [FEV1]) minimizes potential bias arising from the open-label nature of the study. The duration of treatment (12 weeks) was defined based on the guidelines of the Global Initiative for Asthma (GINA 20221) and the Brazilian Society of Pulmonology and Phthisiology (SBPT) regarding the time required to assess the effectiveness of asthma maintenance treatments (three months).

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes who meet all of the following criteria will be included in the study:

* Signature of the Informed Consent Term (ICF) for people over 18 years and, when applicable, signature of the Informed Assent Form (IAF) by the participant under 18 years of age and the ICF by the representative before carrying out any study procedure.
* Age ≥ 12 years.
* History of recurrent symptoms suggestive of asthma (cough, wheezing, shortness of breath, and/or chest tightness).
* Previous medical diagnosis of asthma.

Exclusion Criteria:

Patients who meet at least one of the following criteria will be excluded from the study:

* Occurrence of moderate to serious asthma exacerbation within 90 days prior to initiation of study treatment.
* Presence of acute or chronic symptomatic respiratory tract infection.
* Body mass index (BMI) ≥ 38 kg/m2.
* Use of long-acting anticholinergic drug (LAMA) in the last six (06) months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Absolute change in pre-bronchodilator Forced expiratory volume in one second - Liter, assessed by means of pulmonary function testing 12 weeks after initiation of treatment (Final visit) from baseline (Randomization visit) | of pulmonary function testing 12 weeks after initiation of treatment (Final visit) from baseline (Randomization visit).
  Absolute change in pre-bronchodilator Forced expiratory volume in one second - Liter, assessed by means of pulmonary function testing 12 weeks after initiation of treatment (Final visit) from baseline (Randomization visit). The interval between visits is 28 ± 2 days.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints - treatment progress | Evolution of the pre-bronchodilator Forced expiratory volume in one second - Liter value throughout the treatment (Randomization visit, Visit 1, Visit 2, and Final visit);
  Evolution of the pre-bronchodilator Forced expiratory volume in one second - Liter value throughout the treatment (Randomization visit, Visit 1, Visit 2, and Final visit).The interval between visits is 28 ± 2 days.
Secondary Efficacy Endpoints - treatment progress | Peak expiratory flow value (Liter/minute) measured in the morning and in the afternoon throughout the treatment (Randomization visit, Visit 1, Visit 2, and Final visit);
  Peak expiratory flow value (Liter/minute) measured in the morning and in the afternoon throughout the treatment (Randomization visit, Visit 1, Visit 2, and Final visit).The interval between visits is 28 ± 2 days.
Secondary Efficacy Endpoints - treatment progress | Final Asthma Control Questionnaire 7 score 12 weeks after starting treatment (Randomization visit, Visit 1, Visit 2, and Final visit)
  Final Asthma Control Questionnaire 7 score 12 weeks after starting treatment (Randomization visit, Visit 1, Visit 2, and Final visit).The interval between visits is 28 ± 2 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, Brazil